CLINICAL TRIAL: NCT04146961
Title: The PanOptix Trifocal IOL: A Study of Patient Satisfaction, Visual Disturbances, and Uncorrected Visual Performance
Status: Completed | Type: Observational
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: ALC51819219
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-01

CONDITIONS: Cataract Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Device: Alcon PanOptix or PanOptix Toric IOL — Patients who previously underwent cataract surgery with the Alcon PanOptix or PanOptix Toric IOL in both eyes.

SUMMARY:
Prospective survey study of patients who previously underwent cataract surgery with the Alcon PanOptix or PanOptix Toric intraocular lens in both eyes.

DETAILED DESCRIPTION:
This will be an open-label, prospective survey study of patients who previously underwent cataract surgery with the Alcon PanOptix or PanOptix Toric intraocular lens in both eyes, comparing to an existing historical dataset of patient reported outcomes with bilateral ReSTOR 3.0 implants.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with the PanOptix or Panoptix Toric lenses bilaterally within 6 months of the survey administration. Patients may have the toric version of this lens in neither eye, one eye, or both eyes.
* Patients with otherwise healthy eyes, not exhibiting any significant ocular morbidity that would be expected to influence outcome measures.
* Patients whose spherical equivalent outcome is within 0.5D of target and whose magnitude of manifest postoperative cylinder is less than or equal to 0.75 diopters.

Exclusion Criteria:

* Patients with visually significant co-morbidities (corneal, retina, optic nerve disease) that could affect their satisfaction with surgery.
* Patients with surgical complications either during or after surgery (capsule tears, iris trauma, decentered intraocular lens, cystoid macular edema, etc.)
* Patients with greater than grade 1 posterior capsule opacity.
* Patient sin the historical reference set who underwent Astigmatic Keratotomy or Limbal Relaxing Incision during cataract surgery. -

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The Investigators will collect patient-reported outcomes data on 60 new patients where both eyes receive either a PanOptix or PanOptix Toric lens, depending on the correction needed for each eye to eliminate astigmatism and achieve the target refraction. Both eyes will be targeted for emmetropia. Patients will be screened based on their candidacy for a multifocal implant.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Satisfaction, measured as the percentage of patients reporting "top box" satisfaction | 6/1/20 - 7/1/20
  Primary objective: to determine the percentage of patients who report "top box" (5 out of 5) overall satisfaction on the questionnaire instrument. To determine the percentage of patients who report satisfaction ("satisfied" or "very satisfied" as 4 out of 5 on the attached questionnaire instrument.

SECONDARY OUTCOMES:
Percentage of postoperative patients who report overall satisfaction as either "satisfied" or "very satisfied." | 6/1/20 - 7/1/20
  To report spectacle independence, measured as the percentage of patients who do not require glasses for each of the common activities queried like driving, reading, computer work, watching TV, and sports/hobbies. To determine the incidence of glare and halos described by the patient as "a fair amount" or worse (Question 20).

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, MD, Study Director — Research Insight LLC
Locations (3):
- United States (3):
  - Harvard Eye Associates, Laguna Hills, California
  - Quentin Allen, Palm City, Florida
  - Quantum Vision Center, Edwardsville, Illinois